CLINICAL TRIAL: NCT07153016
Title: LEgal Guidance and AdvocaCY for CAREgivers (LEGACY CARE): A Pilot Clinical Trial for Caregivers of Persons With Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025LS070
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Caregiver Burden; Colorectal Cancer; Legal Intervention
MeSH Terms: conditions — Caregiver Burden; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient - Caregiver Dyads (Experimental): Participants (i.e. patient-caregiver dyads) will receive free, personalized legal care services from Cancer Legal Care (CLC), a nonprofit organization located in the Twin Cities of Minnesota.
  Interventions: Other: Legal Services

INTERVENTIONS:
Other: Legal Services — Legal care services from Cancer Legal Care (CLC), a nonprofit organization located in the Twin Cities of Minnesota.

SUMMARY:
This is a single center single-arm, pilot study of proactive and early connection with free legal care services for patient-caregiver dyads affected by colorectal cancer to assess the feasibility, acceptability, and preliminary efficacy of this intervention in improving financial and psychosocial outcomes.

Participants (i.e. patient-caregiver dyads) will receive free, personalized legal care services from Cancer Legal Care (CLC), a nonprofit organization located in the Twin Cities of Minnesota. The duration of study participation is 3 months, however, participants may continue to access free personalized legal care services beyond this period.

ELIGIBILITY:
Colorectal Cancer Patient Inclusion Criteria:

* Diagnosis of advanced stage (Stage III or Stage IV) colorectal cancer within the past 3 months.
* Initiated or planning to initiate systemic cancer therapy.
* Able to identify a caregiver for study participation.
* Estimated life expectancy of over 6 months in the opinion of the treating oncologist.
* 18 years of age or older at the time of consent.
* Able to understand, speak, read, and write in English.
* Able to provide voluntary written consent prior to the performance of any research related activity.

Caregiver Inclusion Criteria:

* 18 years of age or older at the time of consent.
* Identified as a caregiver by a colorectal cancer patient.
* Able to understand, speak, read, and write in English.
* Able to provide voluntary written consent prior to the performance of any research related activity.

Exclusion Criteria:

* Lacks capacity to consent/diminished capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 3 months
  Feasibility will be measured through rates of 1) initial engagement (i.e., percent of patients and caregivers who meet with a CLC representative), 2) continued engagement (i.e., percentage of patients and caregivers who respond to questionnaires at months 3), and 3) intervention completion (i.e., percentage of patients and caregivers who receive a legal service). The mean of the 3 metrics will be used to determine feasibility. The intervention will be deemed as feasible if ≥50% is met on each of the 3 feasibility metrics.

SECONDARY OUTCOMES:
Acceptability | 3 months
  Acceptability will be assessed through experiences from patients and caregivers. At the end of the 3-months, we will ask all participants how likely they are to recommend this intervention to other patients and/or caregivers (a 5-point Likert scale of likeliness to recommend, ranges from 1-5). 1 meaning the least likely and 5 meaning the most likely to recommend this intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States